CLINICAL TRIAL: NCT02115191
Title: Use of 2-octylcyanoacrylate for Closure Urethrocutaneous Fistulas After Urethroplasty for Hypospadias
Brief Title: 2-octyl Cyanoacrylate for Closure of Urethrocutaneous Fistula.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, GONZALEZ-OJEDA ALEJANDRO, PhD. MD, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Cyanoacrylate-2014-03
Record Dates: First submitted 2014-04-13; First posted 2014-04-15 (Estimated); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Urethrocutaneous Fistulas
Keywords: 2-octylcyanoacrylate; Urethrocutaneous fistulas.; Closure.; Recurrence.
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2-octylcyanoacrylate (Experimental): Application of 2-octylcyanoacrylate
  Interventions: Device: 2-octylcyanoacrylate
- Surgical reintervention (Active Comparator): Surgical reintervention for urethrocutaneous fistula repair
  Interventions: Procedure: Surgical reintervention

INTERVENTIONS:
Device: 2-octylcyanoacrylate — After sedation with midazolam (0.5 mg/kg orally) a Foley catheterization with a 10 Fr gauge siliconized catheter will be placed, with the balloon inflated with 1.5 ml water to prevent bladder spasm. After this we will apply the adhesive by using dissecting forceps to approximate the edges of the UCF, and then apply it several thin layers of OCA.
  Arms: 2-octylcyanoacrylate
Procedure: Surgical reintervention — The reoperation will consist on mobilizing dartos flaps and closing the defect in layers with absorbable sutures. Urinary bladder drainage will be provided with a 10 Fr silicone Foley catheter, with the balloon inflated with 1.5 ml water to prevent bladder spasm.
  Arms: Surgical reintervention

SUMMARY:
Urethrocutaneous fistulae (UCF) represent one of the most frequent causes of morbidity after urethroplasty. Hypospadias can be repaired using different surgical techniques, but regardless of technique, the incidence of UCF ranges between 10% and 40%. The surgical repair of UCF remains the treatment of choice, even if some patients need further operations because of recurrences. The cyanoacrylates have been used as skin suture substitutes, and some evidence suggests a beneficial effect when these adhesives are used as an adjuvant in the management of UCF.

DETAILED DESCRIPTION:
Design Randomized clinical trial carried out in children with UCF that occurred after hypospadias repair. The patients will be assign to either the control or study groups.

The study group will include children with long-standing UCF that occurred at least 6 months after the initial intervention. After preparation of the fistula area, multiple layers of OCA will be apply, attaching the edges of the orifice. The same procedure will be repeated three times and the children will be follow for at least 6 months after treatment.

The control group will include children with long-standing UCF that occurred at least 6 months after the initial intervention. Patients will be scheduled for surgical treatment and will be follow for at least 6 months after surgery. If UCF recurred, a new intervention will be proposed.

The sample size was determined based on a prevalence of the complication (UCF) of 25% in the surgery group and 70% in the medically treated group, given a confidence level of 95% and a power of 0.20, which resulted in a minimum sample size of 18 patients per group.

The independent variables are the application of OCA in the UCF orifice or surgical treatment of UCF and the main outcome variable is FC without recurrence within at least 12 months follow-up. As confounding variables, we considered the children's age, the fistulous orifice diameter and the type of initial surgical procedure to which all were submitted.

Procedure Assignment of patients to groups will be performed by using a sealed envelope chosen randomly by the father, mother or guardians. To decrease the inflammatory response and edema, patients in the study group will be instructed to apply triamcinolone cream to the fistula four times a day for 3 days. Once this treatment is completed, the patient will attended our clinic as an outpatient to undergo, after sedation with midazolam (0.5 mg/kg orally), Foley catheterization with a 10 Fr gauge siliconized catheter, with the balloon inflated with 1.5 ml water to prevent bladder spasm. Subsequently, we will apply an adhesive using dissecting forceps to approximate the edges of the UCF, and then applied several thin layers of OCA.

The urethral catheter will be left in place for 5 days. At the end of this time, we will evaluate the closure or persistence of the UCF. If the UCF persist, the OCA adhesive will be apply twice following the same protocol before the medical procedure was deemed to have failed.

Patients in the control group will wait 6 months to be treated surgically. The reoperation consist on mobilizing dartos flaps and closing the defect in layers with absorbable sutures. Urinary bladder drainage will be provide with a 10 Fr silicone Foley catheter, with the balloon inflated with 1.5 ml water to prevent bladder spasm. The follow-up time will be 12 months for each group.

Statistical analysis Statistical analysis Statistical software, SPSS for IBM (version 20 for Windows; IBM Corp., Armonk, NY, USA) is being used for data analysis.

The data obtained will be expressed as frequencies and percentages, means and standard deviations. For comparing results, Student's t test will be used for continuous variables and Chi2 or Fisher's exact tests will be used for qualitative data when appropriate.

Relative risk (RR) and 95% confidence intervals (95% CI) will be determined as well as the absolute risk reduction (ARR), relative risk reduction (RRR), and number needed to treat (NNT).

Statistical significance from two-tailed tests was assumed when p < 0.05

ELIGIBILITY:
Inclusion Criteria:

* Children younger than 5 years old with at least one postoperative UCF with an external orifice less than 5 mm in diameter at the distal, proximal or medial penis,
* Patients whose parents or guardians accepted inclusion in the study by signing the informed consent form

Exclusion Criteria:

* Patients with an external orifice more than 5 mm in diameter
* Iatrogenic or traumatic fistulae
* The presence of obstruction distal to the fistula, necrotic tissue or active infection at the surgical site,
* The presence of chronic diseases such as diabetes mellitus, renal or hepatic insufficiency, malignancy of any type or use of steroids and/or immunosuppressive therapy of any kind,

Ages: 6 Months to 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2014-04; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Use of 2-octylcyanoacrylate for closure urethrocutaneous fistulas after urethroplasty for hypospadias. | 12 months after procedure.
  Closure or recurrence of urethrocutaneous fistulas after cyanoacrylate application or surgical intervention.

SECONDARY OUTCOMES:
Morbidity after applications | 12 months after the procedure.
  Morbidity after applications of cyanoacrylates or surgical reintervention.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro González-Ojeda, Ph.D., M.D., Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Department of Pediatric Surgery of the Pediatrics Hospital of the Western Medical Center of the Mexican Institute of Social Security, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Derived] Ambriz-Gonzalez G, Aguirre-Ramirez P, Garcia-de Leon JM, Leon-Frutos FJ, Montero-Cruz SA, Trujillo X, Fuentes-Orozco C, Macias-Amezcua MD, del Socorro Alvarez-Villasenor A, Cortes-Flores AO, Chavez-Tostado M, Gonzalez-Ojeda A. 2-octyl cyanoacrylate versus reintervention for closure of urethrocutaneous fistulae after urethroplasty for hypospadias: a randomized controlled trial. BMC Urol. 2014 Nov 21;14:93. doi: 10.1186/1471-2490-14-93. PMID 25416602